CLINICAL TRIAL: NCT05713318
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Assess the Efficacy and Safety of HH-120 Nasal Spray for the Treatment of Mild COVID-19
Brief Title: A Study To Assess The Efficacy and Safety of HH-120 Nasal Spray for the Treatment of Mild COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HH120-NS215
Record Dates: First submitted 2023-01-31; First posted 2023-02-06 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Group 1 (Experimental)
  Interventions: Drug: HH-120 nasal spray
- Treatment Group 2 (Experimental)
  Interventions: Drug: HH-120 nasal spray
- Control Group 3 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator
- Control Group 4 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: HH-120 nasal spray — Nasal spray daily doses of HH-120 4 times added on SOC for 6 consecutive days.
  Arms: Treatment Group 1
Drug: HH-120 nasal spray — Nasal spray daily doses of HH-120 8 times added on SOC for 6 consecutive days.
  Arms: Treatment Group 2
Drug: Placebo Comparator — Nasal spray daily doses of placebo 4 times added on SOC for 6 consecutive days.
  Arms: Control Group 3
Drug: Placebo Comparator — Nasal spray daily doses of placebo 8 times added on SOC for 6 consecutive days.
  Arms: Control Group 4

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 2 study in participants over the age of 18 years with mild COVID-19. The main purpose of this study is to evaluate the effect on viral load clearance and clinical recovery, and safety of HH-120 nasal spray in participants over the age of 18 years with mild COVID-19 (according to the FDA definition, 2021).

ELIGIBILITY:
Inclusion Criteria:

* Participants who are ≥18 years of age .
* Participants who are diagnosed with mild COVID-19 and with Laboratory confirmed of SARS-CoV-2 infection as determined by PCR or antigen test.
* Participants who agree to use highly effective methods of contraception. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test result.
* Participants who are willing and able to provide written informed consent, or with a legal representative who can provide informed consent.

Exclusion Criteria:

* Have suspected or proven serious disease (cardiovascular, renal, liver systems, etc.), active bacterial, fungal, viral, or other infection (except COVID 19) that in the opinion of the Investigator could constitute a risk when taking the study intervention.
* Bronchial asthma or chronic obstructive pulmonary disease （COPD).
* Urgent or expected need for nasal high-flow oxygen therapy or positive pressure ventilation, invasive mechanical ventilation or Extracorporeal membrane oxygenation(ECMO).
* Have prior use (unless required as rescue medication) of any of the following treatments: COVID 19 investigational or Emergency Use Authorization (EUA) approved treatment, including but not limited to convalescent plasma, mAbs against SARS CoV 2, intravenous immune globulin (IVIG) (any indication), where prior use is defined as the past 30 days or less than 5 half lives of the investigational product (whichever is longer) from Screening.
* History of anaphylaxis or other significant allergy in the opinion of the PI or known allergy or hypersensitivity to any of the components of the study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Changes of viral load compared to the baseline | From baseline to Day 7

SECONDARY OUTCOMES:
Time to sustained clinical recovery of 11 COVID-19 symptoms. | From baseline till Day 28
Changes of viral load compared to the baseline. | From baseline till Day 28
Proportion of participants with moderate, severe, critical COVID-19 disease or death. | From baseline till Day 28
Safety assessment: including adverse events, serious adverse events (SAEs), laboratory assessments, etc. | From baseline till Day 28

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou, Fujian
  - The People's Hospital of Gaozhou, Gaozhou, Guangdong
  - Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Lianyungang Oriental Hospital, Lianyungang, Jiangsu
  - Yixing People's Hospital, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Panjin Liaoyou Gem flower Hospital, Panjin, Liaoning
  - Linfen Central Hospital, Linfen, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Qujing First People's Hospital, Qujing, Yunan
  - Southern Central Hospital Of Yunnan Province(The First People's Hospital Of Honghe State), Yisa, Yunnan
  - Wenzhou Traditional Chinese Medicine Hospital, Wenzhou, Zhejiang